CLINICAL TRIAL: NCT02381704
Title: Cost Analysis of Bariatric Surgery in an Employee-based Healthcare System
Brief Title: Cost Analysis of Bariatric Surgery in an Employee-based Healthcare System Following Surgery Coverage
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Dr. Keith Kim, Director of Metabolic Medicine & Surgery Institute at Celebration Health, AdventHealth
Other Study IDs: 08.03.08
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall purpose of the study is to determine prospectively the cost effectiveness of bariatric surgery following partial coverage by a large healthcare system.

DETAILED DESCRIPTION:
Epidemiological studies show that the incidence of morbid obesity is increasing at a considerably greater rate than any other obesity category. The National Institutes of Health, along with a number of medical and scientific national and international professional organizations, recognize that bariatric surgery is the only long-term effective treatment for individuals with morbid obesity. Along with massive and sustained weight loss, bariatric surgery resolves/improves obesity co-morbidities (type 2 diabetes, hypertension, cardiovascular disease, fatty liver disease, asthma, osteoarthritis, fatty liver disease, obstructive sleep apnea, dyslipidemia, hyperlipidemia, infertility, depression, cancer risk, fertility, and more) and significantly increases longevity.

Despite the well-documented benefits of bariatric surgery in terms of health and healthcare costs, many insurers deny coverage for the surgery out of fear that the cost of surgery will financially burden the system. These insurers, however, fail to consider the improvement in obesity-related diseases and associated cost savings. The recent change in policy by the Florida Hospital Healthcare System (FHHS) that allows for partial coverage of bariatric surgery provides the unique opportunity to study prospectively the cost effectiveness of the surgery, i.e. cost of surgery vs. cost savings. Study participants will include approximately 75 to 100 FHHS covered individuals (18 to 64 years) who have been approved for bariatric surgery and who have provided their written consent for study participation.

The study protocol will include a review of patient insurance records for cost analysis of medication and medical expenses prior to surgery and over a two-year period postoperatively. Patients will also be asked to consent to the completion of a yearly questionnaire concerning the status of their obesity co-morbidities, medication use and dosage, and sick leave. The outcome of this prospective study will allow for assessment of the costs of surgery, cost saving in terms of medication and medical expenses, and the potential time period required for return on investment. Such data, when shared with others through peer-review journal publications, may assist other employee healthcare systems in their decision to provide coverage for bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

* Insured under the FHHS
* Have been approved for bariatric surgery
* Have provided their written consent for study participation.

Exclusion Criteria:

* Approved bariatric surgery patients covered by (FHHS)Florida Hospital Healthcare Systems will be excluded from the study if they fail to provide written consent.
* Surgery exclusion:

BMI less than or equal to 35 without at least two major co-morbidities pregnancy active alcoholism or drug abuse suicidal ideation cancer or another wasting disease mental handicap and inability to provide written consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study subjects will include any individual having been approved for surgery that consents to the review of their records and additional survey information pertaining to medication use, dosage, anthropometrics and medical-related days taken. Study subjects would include male and female gender, all ethnicities, ages 18 to 65 years, and exclude populations who do not meet the criteria for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in FHHS expenses pertaining to medical costs incurred by all study participants, as well as those study participants who, prior to their surgery, ranked in the (upper 50th. percentile) vs. (lower 50th. percentile) healthcare utilizing tiers. | one to two years postop

SECONDARY OUTCOMES:
Determine changes in the cost of obesity-related co-morbidities for all study participants and those who, prior to surgery, were within high or low healthcare utilizing tiers. | At the end of postoperative year 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Keith C Kim, MD, Principal Investigator — Advanced Minimally Invasive and Bariatric Surgery Consultants
Locations (1):
- Advanced Minmially Invasive and Bariatric Surgery Consultants, Celebration, Florida, United States

REFERENCES:
- [Background] Seidell JC. Obesity, insulin resistance and diabetes--a worldwide epidemic. Br J Nutr. 2000 Mar;83 Suppl 1:S5-8. doi: 10.1017/s000711450000088x. PMID 10889785
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Freedman DS, Khan LK, Serdula MK, Galuska DA, Dietz WH. Trends and correlates of class 3 obesity in the United States from 1990 through 2000. JAMA. 2002 Oct 9;288(14):1758-61. doi: 10.1001/jama.288.14.1758. PMID 12365960
- [Background] Mokdad AH, Serdula MK, Dietz WH, Bowman BA, Marks JS, Koplan JP. The spread of the obesity epidemic in the United States, 1991-1998. JAMA. 1999 Oct 27;282(16):1519-22. doi: 10.1001/jama.282.16.1519. PMID 10546690
- [Background] Calle EE, Thun MJ, Petrelli JM, Rodriguez C, Heath CW Jr. Body-mass index and mortality in a prospective cohort of U.S. adults. N Engl J Med. 1999 Oct 7;341(15):1097-105. doi: 10.1056/NEJM199910073411501. PMID 10511607
- [Background] Drenick EJ, Bale GS, Seltzer F, Johnson DG. Excessive mortality and causes of death in morbidly obese men. JAMA. 1980 Feb 1;243(5):443-5. PMID 7351764
- [Background] McGee DL; Diverse Populations Collaboration. Body mass index and mortality: a meta-analysis based on person-level data from twenty-six observational studies. Ann Epidemiol. 2005 Feb;15(2):87-97. doi: 10.1016/j.annepidem.2004.05.012. PMID 15652713
- [Background] Sjostrom LV. Mortality of severely obese subjects. Am J Clin Nutr. 1992 Feb;55(2 Suppl):516S-523S. doi: 10.1093/ajcn/55.2.516s. PMID 1531097
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Maggard MA, Shugarman LR, Suttorp M, Maglione M, Sugerman HJ, Livingston EH, Nguyen NT, Li Z, Mojica WA, Hilton L, Rhodes S, Morton SC, Shekelle PG. Meta-analysis: surgical treatment of obesity. Ann Intern Med. 2005 Apr 5;142(7):547-59. doi: 10.7326/0003-4819-142-7-200504050-00013. PMID 15809466
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Kushner RF, Noble CA. Long-term outcome of bariatric surgery: an interim analysis. Mayo Clin Proc. 2006 Oct;81(10 Suppl):S46-51. doi: 10.1016/s0025-6196(11)61180-4. PMID 17036578
- [Background] O'Brien PE, McPhail T, Chaston TB, Dixon JB. Systematic review of medium-term weight loss after bariatric operations. Obes Surg. 2006 Aug;16(8):1032-40. doi: 10.1381/096089206778026316. PMID 16901357
- [Background] Sugerman HJ. Bariatric surgery for severe obesity. J Assoc Acad Minor Phys. 2001 Jul;12(3):129-36. PMID 11851201
- [Background] Martin LF, Lundberg AP, Juneau F, Raum WJ, Hartman SJ. A description of morbidly obese state employees requesting a bariatric operation. Surgery. 2005 Oct;138(4):690-700; discussion 700. doi: 10.1016/j.surg.2005.06.050. PMID 16269298
- [Background] Finkelstein EA, Brown DS. A cost-benefit simulation model of coverage for bariatric surgery among full-time employees. Am J Manag Care. 2005 Oct;11(10):641-6. PMID 16232005
- [Background] Scheen AJ, Letiexhe M, Rorive M, De Flines J, Luyckx FH, Desaive C. [Bariatric surgery: 10-year results of the Swedish Obese Subjects Study]. Rev Med Liege. 2005 Feb;60(2):121-5. French. PMID 15819376
- [Background] Long SD, O'Brien K, MacDonald KG Jr, Leggett-Frazier N, Swanson MS, Pories WJ, Caro JF. Weight loss in severely obese subjects prevents the progression of impaired glucose tolerance to type II diabetes. A longitudinal interventional study. Diabetes Care. 1994 May;17(5):372-5. doi: 10.2337/diacare.17.5.372. PMID 8062602
- [Background] MacDonald KG Jr, Long SD, Swanson MS, Brown BM, Morris P, Dohm GL, Pories WJ. The gastric bypass operation reduces the progression and mortality of non-insulin-dependent diabetes mellitus. J Gastrointest Surg. 1997 May-Jun;1(3):213-20; discussion 220. doi: 10.1016/s1091-255x(97)80112-6. PMID 9834350
- [Background] Malone M, Alger-Mayer SA. Medication use patterns after gastric bypass surgery for weight management. Ann Pharmacother. 2005 Apr;39(4):637-42. doi: 10.1345/aph.1E393. Epub 2005 Mar 1. PMID 15741419
- [Background] Monk JS Jr, Dia Nagib N, Stehr W. Pharmaceutical savings after gastric bypass surgery. Obes Surg. 2004 Jan;14(1):13-5. doi: 10.1381/096089204772787220. PMID 14980027
- [Background] Potteiger CE, Paragi PR, Inverso NA, Still C, Reed MJ, Strodel W 3rd, Rogers M, Petrick A. Bariatric surgery: shedding the monetary weight of prescription costs in the managed care arena. Obes Surg. 2004 Jun-Jul;14(6):725-30. doi: 10.1381/0960892041590999. PMID 15318973
- [Background] Gould JC, Garren MJ, Starling JR. Laparoscopic gastric bypass results in decreased prescription medication costs within 6 months. J Gastrointest Surg. 2004 Dec;8(8):983-7. doi: 10.1016/j.gassur.2004.09.042. PMID 15585385
- [Background] Nguyen NT, Varela JE, Sabio A, Naim J, Stamos M, Wilson SE. Reduction in prescription medication costs after laparoscopic gastric bypass. Am Surg. 2006 Oct;72(10):853-6. PMID 17058720
- [Background] Snow LL, Weinstein LS, Hannon JK, Lane DR, Ringold FG, Hansen PA, Pointer MD. The effect of Roux-en-Y gastric bypass on prescription drug costs. Obes Surg. 2004 Sep;14(8):1031-5. doi: 10.1381/0960892041975677. PMID 15479590
- [Background] Fang J. The cost-effectiveness of bariatric surgery. Am J Gastroenterol. 2003 Sep;98(9):2097-8. doi: 10.1111/j.1572-0241.2003.07671.x. PMID 14499794
- [Background] Martin LF, Tan TL, Horn JR, Bixler EO, Kauffman GL, Becker DA, Hunter SM. Comparison of the costs associated with medical and surgical treatment of obesity. Surgery. 1995 Oct;118(4):599-606; discussion 606-7. doi: 10.1016/s0039-6060(05)80024-8. PMID 7570311
- [Background] Sampalis JS, Liberman M, Auger S, Christou NV. The impact of weight reduction surgery on health-care costs in morbidly obese patients. Obes Surg. 2004 Aug;14(7):939-47. doi: 10.1381/0960892041719662. PMID 15329183
- [Background] Gallagher SF, Banasiak M, Gonzalvo JP, Paoli DP, Allwood J, Morris D, Murr MM, Shapiro DH. The impact of bariatric surgery on the Veterans Administration healthcare system: a cost analysis. Obes Surg. 2003 Apr;13(2):245-8. doi: 10.1381/096089203764467144. PMID 12740132
- [Background] Gorman RS, Stern DL, Inclan DV, Presutti RJ, Swain JM, Hentz JG. Outcomes, health status, and medical resource utilization after bariatric surgery. Compr Ther. 2006 Spring;32(1):34-8. doi: 10.1385/comp:32:1:34. PMID 16785580
- [Background] Kuhlmann HW, Falcone RA, Wolf AM. Cost-effective bariatric surgery in Germany today. Obes Surg. 2000 Dec;10(6):549-52. doi: 10.1381/096089200321594156. PMID 11175964
- [Background] Ackroyd R, Mouiel J, Chevallier JM, Daoud F. Cost-effectiveness and budget impact of obesity surgery in patients with type-2 diabetes in three European countries. Obes Surg. 2006 Nov;16(11):1488-503. doi: 10.1381/096089206778870067. PMID 17132416
- [Background] Clegg A, Colquitt J, Sidhu M, Royle P, Walker A. Clinical and cost effectiveness of surgery for morbid obesity: a systematic review and economic evaluation. Int J Obes Relat Metab Disord. 2003 Oct;27(10):1167-77. doi: 10.1038/sj.ijo.0802394. PMID 14513064
- [Background] Avenell A, Broom J, Brown TJ, Poobalan A, Aucott L, Stearns SC, Smith WC, Jung RT, Campbell MK, Grant AM. Systematic review of the long-term effects and economic consequences of treatments for obesity and implications for health improvement. Health Technol Assess. 2004 May;8(21):iii-iv, 1-182. doi: 10.3310/hta8210. PMID 15147610
- [Background] Finkelstein EA, Brown DS, Avidor Y, Takeuchi AH. The role of price, sociodemographic factors, and health in the demand for bariatric surgery. Am J Manag Care. 2005 Oct;11(10):630-7. PMID 16232004
- [Background] Sadhasivam S, Larson CJ, Lambert PJ, Mathiason MA, Kothari SN. Refusals, denials, and patient choice: reasons prospective patients do not undergo bariatric surgery. Surg Obes Relat Dis. 2007 Sep-Oct;3(5):531-5; discussion 535-6. doi: 10.1016/j.soard.2007.07.004. PMID 17903773
- [Background] Nguyen NT, Paya M, Stevens CM, Mavandadi S, Zainabadi K, Wilson SE. The relationship between hospital volume and outcome in bariatric surgery at academic medical centers. Ann Surg. 2004 Oct;240(4):586-93; discussion 593-4. doi: 10.1097/01.sla.0000140752.74893.24. PMID 15383786
- [Background] Murr MM, Martin T, Haines K, Torrella T, Dragotti R, Kandil A, Gallagher SF, Harmsen S. A state-wide review of contemporary outcomes of gastric bypass in Florida: does provider volume impact outcomes? Ann Surg. 2007 May;245(5):699-706. doi: 10.1097/01.sla.0000256392.04141.04. PMID 17457162
- [Result] 6. CDC. Obesity and overweight trends. http://www.cdc.gov/nccdphp/dnpa/obesity/trend/index.htm
- [Result] Brethauer SA, Chand B, Schauer PR. Risks and benefits of bariatric surgery: current evidence. Cleve Clin J Med. 2006 Nov;73(11):993-1007. doi: 10.3949/ccjm.73.11.993. PMID 17128540
- [Result] Buffington CK, Cowan GSM, Jr. Gastric Bypass in the Treatment of Diabetes, Hypertension and Lipid/lipoprotein Abnormalities of the Morbidly Obese. In Deitel M (ed.): Companion Volume to Obesity Surgery for the Morbidly Obese Patient. 2000 by FD Publications, Toronto, Canada, pp. 435-450.
- [Result] North American Association for the Study of Obesity and the National Heart, Lung, and Blood Institute. The practical guide: identification, evaluation and treatment of overweight and obesity in adults. Bethesda, MD. National Institutes of Health, 2000, NIH Publication 00-4084.
- [Result] North American Association for the Study of Obesity and the National Heart, Lung, and Blood Institute. Clinical Guidelines on the identification, evaluation, and treatment of overweight and obesity in adults. The Evidence Report. Bethesda, Md: National Institutes of Health, 1998. NIH Publication 98-4083.
- [Result] Colquitt J, Clegg A, Loveman E, Royle P, Sidhu MK. Surgery for morbid obesity. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD003641. doi: 10.1002/14651858.CD003641.pub2. PMID 16235331